CLINICAL TRIAL: NCT01840813
Title: Intra-umbilical Injection of Misoprostol Versus Normal Saline in the Management of Retained Placenta: Intrapartum Placebo-controlled Trial
Brief Title: Intraumbilical Misoprostol in Retained Placenta
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Assistant Prof. Shahla Alalaf, Assistant Professor, Hawler Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMU911
Record Dates: First submitted 2013-04-18; First posted 2013-04-26 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Retained Placenta
Keywords: Intraumbilical misoprostol; Retained placenta; Active management of third stage of labour
MeSH Terms: conditions — Placenta, Retained | interventions — Misoprostol; Saline Solution

ARMS (2):
- Misoprostol (Active Comparator): 4 misoprostol tablets (Misotac® 200 micrograms tablet) dissolved in 20 ml of normal saline injected to umbilical vein
  Interventions: Drug: Misoprostol
- Normal saline (Placebo Comparator): Normal saline 0.9%, 20 ml was injected in the umbilical vein in cases of retained placenta
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Misoprostol — It is a synthetic prostaglandin (PgE1 analogue)used as a uterotonic substance.
  Other Names: (Misotac)® tablet
  Arms: Misoprostol
Drug: Normal saline — It is a placebo group
  Other Names: Normal saline 0.9%
  Arms: Normal saline

SUMMARY:
Administration of intraumbilical misoprostol to women with retained placenta despite active management of third stage of labour reduces the need for manual removal of placenta and the amount of blood loss vaginally.

DETAILED DESCRIPTION:
Retained placenta (RP)is one of the complications of third stage of labour; it should be managed promptly as it may cause severe bleeding, infection, maternal morbidity and mortality .The current standard management of RP word wide, by manual removal aims to prevent these problems, but it is unsatisfactory method because it requires general anaesthesia in hospital, It is an invasive procedure with its own serious complications of bleeding, infection and genital tract injury. Umbilical vein injection of misoprostol is a simple, safe method and could be performed at the place of delivery .

ELIGIBILITY:
Inclusion Criteria:

* women having singleton pregnancy
* 28 weeks of gestation or more delivered vaginally
* prolongation of the third stage of labour (more than 30 min) following active management of third stage of labour

Exclusion Criteria:

* Who refused to participate in the trial
* Multiple pregnancies
* Previous Caesarean Section
* Haemodynamically unstable
* Severe anaemia (haemoglobin less than 8gm/dl)
* Chorioamnionitis

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2011-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
delivery of placenta by medical intervention | 30 minutes after the injection of misoprostol or normal saline in the umbilical vein
  The administration of intraumbilical misoprostol to women with retained placenta despite active management of third stage of labour reduces the need for manual removal of placenta under general anaesthesia.

SECONDARY OUTCOMES:
vaginal bleeding after misoprostol use | 30 minutes after umbilical vein injection of misoprostol
  using intraumbilical misoprostol in women with retained placenta reduces the amount of blood loss vaginally.

OTHER OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolabrity | 2 hours after umbilical vein injection of misoprostol
  Local applications of misoprostol through umbilical vein is associated with less side effects like shivering, fever, dizziness vomiting, flushes, nausea, abdominal pain and headache

CONTACTS AND LOCATIONS:
Overall Officials: Shahla K. Alalaf, Clinical M.D, Principal Investigator — Hawler Medical University; Sheelan S Rajab, High Diploma, Study Chair — , Shaheed Dr.Khalid General Hospital, Directorate of Health
Locations (1):
- Maternity Teaching Hospital, Erbil, Kurdistan Region, Iraq